CLINICAL TRIAL: NCT00682136
Title: Efficacy of Local Anesthetic TAP Blocks in Providing Pain Relief Following Laparoscopic and Open Abdominal Surgery
Brief Title: Analgesic Efficacy of Local Anesthetic Transversus Abdominis Plane (TAP) Blocks in Abdominal Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hunter Colorectal Research (Other)
Responsible Party: Dr Brian Draganic, Hunter Colerectal Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TAPTRIAL; 08/02/20/3.02
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Pain
Keywords: postoperative analgesia; abdominal surgery; ropivacaine; local anaesthesia; tap block; pain management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Open Laparotomy Arm: All patients enrolled in the study who are undergoing elective open laparotomy surgery.
  Interventions: Procedure: US-Guided Ropivacaine TAP Block
- 2 (Active Comparator): Laparoscopic Arm: All patients enrolled in the study who are undergoing elective laparoscopic abdominal surgery.
  Interventions: Procedure: US-Guided Ropivacaine TAP Block

INTERVENTIONS:
Procedure: US-Guided Ropivacaine TAP Block — Bilateral injection of local anaesthetic into the Transversus Abdominis plane, guided by ultrasound.
  Other Names: TAP Block

SUMMARY:
The aim of the study is to establish the efficacy of local anaesthetic TAP (transversus abdominis plane) blocks in providing pain relief in the first 24hrs following open or laparoscopic elective abdominal colorectal operations.

TAP blocks involve the injection of local aesthetic (ropivicaine) into the transversus abdominis plane in the abdominal wall. This injection takes place after induction of anaesthesia, but before the commencement of surgery. TAP blocks have been proposed as a potential safer alternative to epidural anaesthesia. The blocks have been extensively used in the Hunter New England system over the last 18 months. As yet there is no clear evidence for there efficacy, hence the need for this trial.

This trial would establish the efficacy of this practice. If the technique proves effective it could be widely used and provide a simpler method of managing post operative pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and over undergoing elective open or laparoscopic colorectal surgery performed by the participating surgeons within the study period will be considered for the trial.

Exclusion Criteria:

* History of adverse reaction to Ropivicaine or similar drug.
* Inability or refusal to give consent
* Coagulopathic
* Severe renal impairment
* Aged <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
mg/kg of morphine equivalent used by patients post operatively. | From operation until discharge.

SECONDARY OUTCOMES:
Lung Function (spirometry), including FVC, FEV1 and PEFR | 24, 48 and 72 hours postoperatively
Visual Analogue Scale for pain at rest, deep breathing and coughing. | 24, 48 and 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Brian Draganic, B.Med.,B.Med.Sci.(Hons),FRACS, Principal Investigator — Hunter Colorectal Research; Stephen Smith, B.Med.,F.R.A.C.S., Principal Investigator — Hunter Colorectal Research
Locations (4):
- Australia (4):
  - John Hunter Hospital, New Lambton, New South Wales
  - Newcastle Private Hospital, New Lambton, New South Wales
  - Private Medical Suites, New Lambton, New South Wales
  - Mater Misericordiae Hospital, Waratah, New South Wales